CLINICAL TRIAL: NCT06180668
Title: Global Outcomes After Laparotomy for Trauma: The GOAL-Trauma Study
Brief Title: Global Outcomes After Laparotomy for Trauma
Acronym: GOAL-Trauma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Michael Bath, Research Student, University of Cambridge
Other Study IDs: GlobalTraumaLaprotomy
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Abdominal Trauma
MeSH Terms: conditions — Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trauma Laparotomy Patients: Patients of all ages who present to hospital with a blunt or penetrating injury and undergo a trauma laparotomy within 5 days of presentation to the treating centre
  Interventions: Procedure: Trauma Laparotomy

INTERVENTIONS:
Procedure: Trauma Laparotomy — Emergency abdominal surgery through midline incision to access abdominal and / or pelvic organs, to access identified injuries or exploratory diagnostic reasons

SUMMARY:
The goal of this observational study is to assessing the global variation in patient characteristics, management, and outcomes in those undergoing trauma laparotomy.

The main questions it aims to answer are:

* What are the post-operative mortality rates for patients undergoing a trauma laparotomy globally
* What are the epidemiological characteristics (demographics, injury characteristics, baseline clinical characteristics, and surgical case mix) for patients undergoing a trauma laparotomy
* What are the pre-operative, peri-operative, and post-operative processes of care for patients undergoing a trauma laparotomy

This is a purely observational study on patients undergoing trauma laparotomy, with no direct change to clinical care.

DETAILED DESCRIPTION:
We will conduct a prospective multi-centre observational cohort study of patients undergoing a trauma laparotomy. We will recruit centres through pre-existing research networks, utilising a snowballing technique to expand registration of centres. We will enrol eligible patients undergoing emergency trauma laparotomy over a consecutive 30 day period at individual centres during the study dates, with patients followed until discharge, death, or 30 days post-operatively, whichever comes first. All data will be submitted to a central study team by 30 days after the end of their respective data study period.

Any hospital worldwide that performs emergency trauma surgery will be eligible to participate, including both trauma centres and trauma units; a minimum of 1 case must be submitted by the centre during the 30 day study period to be eligible. Each centre's team will be comprised of a local study lead, with maximum 3 members of the local study team for each data collection period. Independent data validators will be also required for select centres.

We will include patients of all ages who present to hospital with a blunt or penetrating injury and undergo a trauma laparotomy within 5 days of presentation to the treating centre (day 0 being time of presentation). A patient will be included for final analysis if >70% of the data points required have been recorded.

Exclusion criteria are:

* Patients undergoing a laparotomy ≥ 5 days (i.e. 120 hours) since presentation to the treating centre
* Any relook laparotomy, including transfers from another centre for further and / or definitive surgery
* Any laparoscopic (including laparoscopic converted to open), robotic, or image-guided procedures
* Patients who have been recently discharged from any hospital (including for non-trauma related admissions) and have represented within 30 days of discharge

We aim to collect system, patient, process, and outcome data. A data set will be collected on all patients undergoing a trauma laparotomy within the inclusion period. The included data fields were based on work by similar studies and refined through iterative consultation with a global interdisciplinary consortium of clinicians involved in trauma care.

Data will be collected through access to patient records only at each centre, performed by members of the local study team. The patient will not be contacted directly in any capacity during their inpatient stay or after the study and no direct involvement in patient care will occur. Data will be collected directly onto a well-established secure web-based system, REDCap cloud (or recorded temporarily onto a hard copy Data Collection Form and uploaded to REDCap at a later date)

The data collected will include a pragmatic set of variables that allow the proposed research to be conducted, but minimise both risk of identification and exclude extraneous possibly sensitive medical information. Local requisite ethics and approvals will be applied for and be in place before any data collection occurs.

ELIGIBILITY:
Inclusion Criteria:

* Any patients of any ages who presents to hospital with a blunt or penetrating injury and undergo a trauma laparotomy within 5 days of presentation to the treating centre

Exclusion Criteria:

* Patients undergoing a laparotomy ≥ 5 days (i.e. 120 hours) since presentation to the treating centre
* Any relook laparotomy, including transfers from another centre for further and / or definitive surgery
* Any laparoscopic (including laparoscopic converted to open), robotic, or image-guided procedures
* Patients who have been recently discharged from any hospital (including for non-trauma related admissions) and have represented within 30 days of discharge

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing a trauma laparotomy for either a blunt or penetrating injury within 5 days of presenting to the treating centre.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days post-operatively
  All cause 30-day post-operative mortality rate

SECONDARY OUTCOMES:
Length of Hospital Stay | 30 days post-operatively
  Time in hospital, from the operation until discharge
Morbidity Rates | 30 days post-operatively
  Any post-operative morbidity that occurred to the patient, as defined by the adapted Clavien-Dindo in trauma scale
Discharge Destination | 30 days post-operatively
  At time of discharge or stepdown from hospital, location the patient was discharged

CONTACTS AND LOCATIONS:
Overall Officials: Tom Bashford, PhD, Principal Investigator — University of Cambridge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bath MF, Amoako J, Kohler K, Hashi AS, Zhang Z, Baderhabusha DU, Caceres E, Nuno-Guzman CM, Marsden M, Carenzo L, Khajanchi M, Saleh R, Edmiston T, Hammer C, Hobbs L, Smith BG, Hutchinson P, Weiser TG, Perkins ZB, Hardcastle TC, Bashford T; GOAL-Trauma Collaborative. Global variation in patient factors, interventions, and postoperative outcomes for those undergoing trauma laparotomy: an international, prospective, observational cohort study. Lancet Glob Health. 2025 Nov;13(11):e1837-e1848. doi: 10.1016/S2214-109X(25)00303-1. Epub 2025 Sep 16. PMID 40972623
- See also: Main Study Website — https://goaltrauma.org/